CLINICAL TRIAL: NCT01583920
Title: Pilot Study of Focal Salvage HDR Prostate Brachytherapy
Brief Title: Focal Salvage HDR Brachytherapy for the Treatment of Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry)
Responsible Party: Principal Investigator, Dr. Hans Chung, Dr. Hans Chung, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: clinicaltrials_hchu_042012
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: prostatic neoplasms; brachytherapy; salvage therapy; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal salvage HDR prostate brachytherapy (Experimental)
  Interventions: Radiation: focal salvage HDR prostate brachytherapy

INTERVENTIONS:
Radiation: focal salvage HDR prostate brachytherapy — Treatment will be delivered using 192-Ir HDR afterloading. Dose prescription is 2 fractions of 13.5 Gy each, delivered 1 week apart.

SUMMARY:
Radiation therapy is considered a standard treatment option for the management of localized prostate cancer. Among the 20-30% who recur, a proportion of them will present with an isolated local recurrence, meaning no distant metastases. If left untreated, it may serve as a source for subsequent metastases. Salvage options available for isolated local recurrence include; temporary or permanent implantation of radioactive seeds into the prostate, complete removal of the prostate gland, use of low temperatures to treat the disease, and high frequency ultrasound to treat the disease. There are risks of complications associated with all these treatments, and there is presently no consensus as to which treatment is the best. Therefore, the aim of this pilot study is to look at the feasibility and toxicities of focal treatment of the prostate using temporary implantation of radioactive seeds into the prostate which the investigators hope will be less since the entire prostate is not treated.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed locally recurrent prostate adenocarcinoma > 30months after the completion of XRT, SBRT, LDR or HDR brachytherapy boost with XRT, or LDR or HDR brachytherapy as monotherapy by a stereotactic transperineal biopsy
* Staging T2-weighted, DWI and DCE-MRI that demonstrates solitary recurrence confined to prostate, and correlates with stereotactic transperineal biopsy
* Staging CT or MRI (abdomen and pelvis) and bone scan are negative for metastases
* American Urological Association Symptom Index Score (ie. IPSS) < 15
* Baseline (post-XRT) serum PSA < 10 ng/mL
* Prostate volume as measured by transrectal ultrasound (TRUS) < 50cc
* ECOG performance status 0-1

Exclusion Criteria:

* Any of the following prior therapies: transurethral resection of the prostate (TURP), radionuclide (permanent or temporary implantation) prostate brachytherapy, prostatectomy or prostatic cryosurgery, HIFU (high-intensity focused ultrasound), bilateral orchiectomy, chemotherapy for prostatic carcinoma
* Evidence of castrate resistance (defined as PSA > 3 ng/mL while testosterone is < 1.7 nmol/L). Patients could have been on combined androgen blockade with initial radiotherapy but are excluded if this was started due to PSA progression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute urinary and rectal toxicities | Acute period (<6 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v4.0

SECONDARY OUTCOMES:
Incidence of late urinary and rectal toxicities | Late period (>6 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Biochemical (ie. prostate specific antigen) disease free survival | 5 years
Quality of Life (QoL) | 5 years
  Expanded Prostate Cancer Index Composite (EPIC)
Acute and late urinary toxicities | 5 years
  American Urological Association Symptom Index Score (i.e. IPSS)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Chung, MD, Principal Investigator — Sunnybrook Health Sciences Centre, Odette Cancer Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Paulin G, Morton G, Loblaw A, Tseng CL, Corkum M, Murgic J, Ravi A, Davidson M, Wronski M, Paudel M, Haider M, Deabreu A, Zhang L, Chung HT. Updated results of MR-assisted focal salvage HDR prostate brachytherapy: a prospective study. Radiother Oncol. 2025 Oct;211:111091. doi: 10.1016/j.radonc.2025.111091. Epub 2025 Aug 9. PMID 40789422